CLINICAL TRIAL: NCT01010516
Title: Comparison of High-Dose Rosuvastatin Versus Low Statin Dose Plus Fenofibrate Versus Low Statin Dose Plus Niacin in the Treatment of Mixed Hyperlipidemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ioannina (Other)
Responsible Party: Prof Moses Elisaf, University of Ioannina Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2009-11

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-dose rosuvastatin (Active Comparator): 40 mg of rosuvastatin
  Interventions: Drug: High-dose rosuvastatin
- Stain plus fenofibrate (Active Comparator): existing statin plus micronized fenofibrate 200 mg
  Interventions: Drug: Statin plus fenofibrate
- Statin plus niacin ER/laropiprant (Active Comparator): existing statin plus extended-release niacin/laropiprant (1 g/day for the first month which will be uptitrated to 2 g/day for the next months)
  Interventions: Drug: Statin plus niacin ER/laropiprant

INTERVENTIONS:
Drug: High-dose rosuvastatin — 40 of rosuvastatin daily
  Arms: High-dose rosuvastatin
Drug: Statin plus fenofibrate — Existing statin plus micronised fenofibrate 200 mg daily
  Arms: Stain plus fenofibrate
Drug: Statin plus niacin ER/laropiprant — Existing statin plus extended-release niacin/laropiprant (1 g/day for the first month which will be uptitrated to 2 g/day for the next months)
  Arms: Statin plus niacin ER/laropiprant

SUMMARY:
Statin therapy does not fully eliminate the cardiovascular disease (CVD) risk associated with low high density lipoprotein-C (HDL-C) and high triglyceride levels. It is currently unknown what would be the best treatment option for patients with mixed hyperlipidemia who fail to meet their lipid targets with statin monotherapy at conventional does, i.e. high dose rosuvastatin or conventional statin dose plus micronized fenofibrate or conventional statin dose plus niacin/laropiprant. The aim of the present study is to compare the efficacy of high-dose rosuvastatin vs conventional statin dose plus micronized fenofibrate vs conventional statin dose plus extended-release niacin/laropiprant on lipid profile in patients with mixed hyperlipidemia. The primary efficacy endpoint will be changes in non-HDL-C levels at 6 months after treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Non-HDL-C above target goal according to NCEP-ATP III after 3 months of treatment with conventional statin doses, e.g. simvastatin 10-40 mg, atorvastatin 10-40 mg or rosuvastatin 5-20 mg

Exclusion Criteria:

* Known CVD, triglycerides > 500 mg/dL, renal disease (serum creatinine levels > 1.6 mg/dL), hypothyroidism [thyroid stimulating hormone (TSH) > 5 IU/mL], liver disease (ALT and/or AST levels > 3-fold upper limit of normal in more than 2 consecutive measurements), alcohol consumption > 3 drinks/day for men and > 2 drinks/day for women, and current or previous gout.
* Patients with diabetes will be included in the study if they are adequately controlled (HbA1c <7%) with one or 2 antidiabetic drugs (no change in their treatment will be made during the study period).
* Patients with hypertension will be included in the study if they are on stable medication for at least 3 months and their blood pressure is adequately controlled (no change in their treatment will be made during the study period).
* Patients currently taking lipid-lowering drugs (other than statins at a conventional dose) or having stopped them less than 4 weeks before study entry will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Changes in non-HDL-C levels | 6 months after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Moses S Elisaf, MD, Principal Investigator — University of Ioannina Medical School
Locations (1):
- University of Ioannina Medical School, Ioannina, Greece

REFERENCES:
- [Derived] Kei A, Tellis C, Liberopoulos E, Tselepis A, Elisaf M. Effect of switch to the highest dose of rosuvastatin versus add-on-statin fenofibrate versus add-on-statin nicotinic acid/laropiprant on oxidative stress markers in patients with mixed dyslipidemia. Cardiovasc Ther. 2014 Aug;32(4):139-46. doi: 10.1111/1755-5922.12072. PMID 24618208
- [Derived] Kei A, Liberopoulos E, Elisaf M. Effect of hypolipidemic treatment on glycemic profile in patients with mixed dyslipidemia. World J Diabetes. 2013 Dec 15;4(6):365-71. doi: 10.4239/wjd.v4.i6.365. PMID 24379928
- [Derived] Kei A, Liberopoulos E, Tellis K, Rizzo M, Elisaf M, Tselepis A. Effect of hypolipidemic treatment on emerging risk factors in mixed dyslipidemia: a randomized pilot trial. Eur J Clin Invest. 2013 Jul;43(7):698-707. doi: 10.1111/eci.12095. Epub 2013 Apr 20. PMID 23600368
- See also: 2nd Department of Internal Medicine, University Hospital of Ioannina — http://www.bpath.gr
- See also: University of Ioannina. Greece — http://www.uoi.gr
- See also: University Hospital of Ioannina, Greece — http://www.uhi.gr